CLINICAL TRIAL: NCT05597618
Title: Evaluation of the Effectiveness of the Training Program Developed to Empower New Graduated Nurses
Brief Title: Empowerment Program for New Graduated Nurses
Acronym: Empowerment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Sevilay Senol Celik, Professor, Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: secelik
Record Dates: First submitted 2022-10-18; First posted 2022-10-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Empowerment
Keywords: Education; Empowerment; Graduated; Nurses; Training
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Intervention Model Description: Sixty-eight participants were randomly selected from the list of newly graduated nurses from the hospital using a simple random numbers table. After obtaining consent from the participants and evaluating the inclusion criteria, 68 participants were randomly assigned to the experimental and control groups. Using the block randomization method (randomizer.org), these nurses were assigned to the experimental and control groups by a research assistant in the institution where the researchers were not involved in the study work.
Who Masked: Participant, Outcomes Assessor
Masking Description: The masking technique was used in the randomization process in the research, and care was taken not to know who was in the intervention and who was in the control group during the assignment process until the study started. In the process of hiding random assignment, the closed envelope method was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervantion Group (No Intervention): Application Steps of Control Group New Graduated Nurses The control group nurses will be required to fill in the "Introductory Information Questionnaire, Empowerment Information Evaluation Questionnaire, Nursing Structural Empowerment Scale, and Psychological Empowerment Scale" in the randomization process.
- Experimental Group (Experimental): Application Steps of Experimental Group New Graduated Nurses In the first stage, the experimental group nurses will be required to fill in the "Introductory Information Questionnaire, Information Evaluation Questionnaire for Empowerment, Nursing Structural Empowerment Scale, and Psychological Empowerment Scale" in the randomization process.
  In the second stage, the theoretical part of the training program will be given to nurses as group training in a physical environment. After the training, the first part of the Training Evaluation Form and the Empowerment Information Evaluation Questionnaire will be applied.
  In the third stage, nurses will be required to use the developed mobile-compatible online training program for 6 months.
  In the fourth stage, Education Evaluation Form, the Nursing Structural Empowerment Scale, the Psychological Empowerment Scale, and the Empowerment Information Evaluation Questionnaire will be applied to the nurses after 6 months.
  Interventions: Other: Training Program to be Developed for Empowering New Graduated Nurses

INTERVENTIONS:
Other: Training Program to be Developed for Empowering New Graduated Nurses — The training program, which will be prepared based on structural and psychological empowerment theories, will consist of two parts: face-to-face theoretical training and online training.
  1. Theoretical Education Part In the theoretical part, empowerment based on structural and psychological empowerment theories, effective communication, problem-solving and decision-making, time management, stress management, and nursing legislation will occur. In addition, the subject related to the institution's promotion (organizational chart, vision, mission, values, etc.) will be included.
  2. Online Education Part In the online part; Videos of theoretical education subjects, institutional information, and documents (institutional instructions and procedures, institution vision-mission-values, management chart, etc.), nursing-related legislation (nursing law, nursing regulation), nursing ethical codes and case studies of sample subjects are included.
  Arms: Experimental Group

SUMMARY:
This study aimed to develop a training program for the empowerment of newly graduated nurses and to evaluate the effectiveness of this program. The training program designed to empower newly graduated nurses is based on the theories of "structural empowerment" and "psychological empowerment." The training program consists of two parts: face-to-face theoretical training and online training. To evaluate the effectiveness of the training program to be developed for the empowerment of newly graduated nurses, the research was planned as a single-center, parallel-group randomized controlled study, following the Consolidated Reporting Trials Standards (CONSORT) guidelines. The main questions it aims to answer are:

1. Is there a difference between the structural empowerment perception levels of the experimental group nurses who received the empowerment training program and the control group nurses who went through the routine orientation program?
2. Is there a difference between the psychological empowerment perception levels of the experimental group nurses who received the empowerment training program and the control group nurses who went through the routine orientation program? The research population will be newly graduated nurses (12 months or less of experience) working at Koç University Hospital. Experimental and control groups are expected to apply questionnaires including the "Introductory Information Questionnaire, Empowerment Information Evaluation Questionnaire, Nursing Structural Empowerment Scale, and Psychological Empowerment Scale" as a pre-test. Nurses in the control and experimental groups will receive the routine practices of the institution. The training program developed in addition to the experimental group will be applied. Six months after the training, the experimental and control groups are expected to apply the questionnaires, including the Nursing Structural Empowerment Scale, the Psychological Empowerment Scale, and the Empowerment Information Evaluation Questionnaire as a post-test.

DETAILED DESCRIPTION:
It is known that newly graduated nurses are influential in individual, institutional, and patient outcomes and encounter many problems. Most healthcare institutions do not implement a planned adaptation program for newly recruited nurses. These nurses try to adapt to the institution and the profession with a master-apprentice relationship. In some of them, a basic adaptation program limited to a specific period is implemented. However, there is no theory-based, innovative, easy-to-use training program and any mobile application to increase the qualifications of newly graduated nurses, who play an essential role in the delivery and quality of health services, to ensure corporate belonging, and to support and strengthen their professionalization and professional competence. In addition, there is no study on this subject. The mobile application study was planned as a randomized controlled study to evaluate the effectiveness of the training program for the empowerment of newly graduated nurses and the mobile application to be developed. In the creation of the content of the training program, descriptive and qualitative studies aiming at strengthening the situation assessment will be carried out. In the research, "Control and Experimental Group Introductory Information Questionnaire," "Status Evaluation Questionnaire for Empowerment," "Nursing Structural Empowerment Scale," "Psychological Empowerment Scale, "Semi-structured Interview Form for New Graduated Nurses," and "Information Evaluation for Empowerment." "Question Form" and "Education Evaluation Form" will be used. Gpower 3.1.9.6 by taking 90% power, 0.81 effect size, and first type error 0.05 of the study's sample. As a result of the power analysis made with the help of software, It was decided to have 68 people, 34 in the experimental group and 34 in the control group. Statistical evaluations of the research data will be made using SPSS 26.

ELIGIBILITY:
Inclusion Criteria:

* Total working time in the profession is less than 12 months
* Having at least a bachelor's degree in nursing

Exclusion Criteria:

* Total working time in the profession is over 12 months
* Dismissal during the research process
* Having an education level below the undergraduate level

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Nursing Structural Empowerment Scale | Change from Nursing Structural Empowerment Levels at 6 months
  The Nursing Structural Empowerment Scale, developed based on Kanter's theory, was revised by Laschinger in 2001 and took its final form (CWEQ-II). The scale is used to evaluate nurses' perception of workplace structural empowerment and consists of 6 dimensions and 19 items as access to opportunities, access to information, access to resources, support, and formal and informal power. To obtain construct validity, a 2-item Global Empowerment Sub-Scale was added to the scale in 1995, and this score was not included in the scale score. The structural reinforcement scale is in a 5-point Likert style. The General Reinforcement score is obtained by adding and averaging the two general enhancement items at the end of the questionnaire. The total score between 6-13 indicates low, the total score between 14-22 indicates medium, and the total score between 23-30 indicates a high level of empowerment perception.
Psychological Empowerment Scale | Change from Nursing Psychological Empowerment Levels at 6 months
  The psychological empowerment scale was developed by Spreitzer in 1995. In the scale, psychological empowerment is defined under four dimensions: meaning, competence, autonomy, and impact. There are 12 questions in total, three of which are in each dimension of psychological empowerment in the scale. The questions are in a 7-point Likert type. The scores of the answers given to the statements in the scale are summed to obtain the psychological empowerment score. The lowest score obtained from the scale is 12, which indicates low psychological empowerment perception, while the highest score is 84, which indicates high psychological empowerment perception.

SECONDARY OUTCOMES:
Empowerment Information Evaluation Questionnaire | Change from Empowerment Knowledge Level at 6 months
  This questionnaire contains multiple-choice questions about the subjects in the training program to be applied to the experimental group of the research. It contains 20 questions in total.

CONTACTS AND LOCATIONS:
Overall Officials: Sevilay Şenol Çelik, MSN, Study Director — Koc University School of Nursing
Locations (1):
- Koç University School of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, and informed consent form will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning nine months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Im SB, Cho MK, Kim SY, Heo ML. The Huddling Programme: effects on empowerment, organisational commitment and ego-resilience in clinical nurses - a randomised trial. J Clin Nurs. 2016 May;25(9-10):1377-87. doi: 10.1111/jocn.13228. Epub 2016 Mar 16. PMID 26990685
- [Background] Kuokkanen L, Leino-Kilpi H, Numminen O, Isoaho H, Flinkman M, Meretoja R. Newly graduated nurses' empowerment regarding professional competence and other work-related factors. BMC Nurs. 2016 Mar 24;15:22. doi: 10.1186/s12912-016-0143-9. eCollection 2016. PMID 27013927
- [Background] Spence Laschinger HK, Nosko A, Wilk P, Finegan J. Effects of unit empowerment and perceived support for professional nursing practice on unit effectiveness and individual nurse well-being: a time-lagged study. Int J Nurs Stud. 2014 Dec;51(12):1615-23. doi: 10.1016/j.ijnurstu.2014.04.010. Epub 2014 Apr 19. PMID 24810929
- [Result] Laschinger HK, Finegan J, Shamian J. The impact of workplace empowerment, organizational trust on staff nurses' work satisfaction and organizational commitment. Health Care Manage Rev. 2001 Summer;26(3):7-23. doi: 10.1097/00004010-200107000-00002. PMID 11482178
- [Result] Spreitzer, G. M. Psychological empowerment in the workplace: Dimension, measurement, and validation. The Academy of Management Journal. 1995; 38(5): 1442-1465.